CLINICAL TRIAL: NCT06369415
Title: Long-term Developmental and Behavioral Outcomes of Children Born From CAPA-IVM Versus Conventional IVF at 5-year-old
Brief Title: Health of Babies Born From IVF Versus IVM at 5 Years Old
Acronym: FM-BABIES-5Y
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 04/24/DD-BVMD
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Infertility; IVF; IVM; Development, Child
Keywords: IVF; IVM; ASQ-3; childhood development
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IVM children: Children born from in-vitro maturation.
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 and behavioural screening according to Strength and Difficulties Questionnaires (SDQ's)
- IVF children: Children born from conventiona in-vitro fertilization.
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 and behavioural screening according to Strength and Difficulties Questionnaires (SDQ's)

INTERVENTIONS:
Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 and behavioural screening according to Strength and Difficulties Questionnaires (SDQ's) — Ages & Stages Questionnaires®, Third Edition (ASQ®-3) is a developmental screening tool designed for use by early educators and health care professionals. It relies on parents as experts, is easy to use, family-friendly and creates the snapshot needed to catch delays and celebrate milestones. The ASQ-3 covers five developmental domains: communication, gross motor, fine motor, problem-solving and personal-social behaviour.
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire for 2-17-year-olds. It exists in several versions to meet the needs of researchers, clinicians and educationalists. The SDQ asks about 25 attributes, some positive and others negative. These 25 items are divided between 5 scales: emotional symptoms, conduct problems; hyperactivity/inattention, peer relationship problems, and prosocial behaviour

SUMMARY:
The investigators conduct a long-term follow-up at five years on offspring born from our randomized controlled trial (RCT) to investigate whether or not there is any difference in developmental outcomes in children born after capacitation IVM (CAPA IVM) compared with conventional IVF in order to give strong evidence about the safety of IVM in women with high antral follicle count.

DETAILED DESCRIPTION:
The safety of the CAPA-IVM has also been proven by publications about the development of children born from this technique.

Data monitoring the physical, mental, and motor development of children born from the CAPA-IVM versus children born from the conventional IVF after 2 years under using the ASQ-3 tools and red flags showed that there were no significant differences in ASQ-3 scores at 6, 12 and 24 months between children born after IVM or IVF. The proportion of children with developmental red flags was low and did not differ between the two groups. Slightly, but significantly, lower ASQ-3 problem-solving and personal-social scores in twins from the IVM versus IVF group at 6 months were still within the normal range and had caught up to the IVF group in the 12- and 24-month assessments.

However, another question raised is whether there is a difference in the development of children born from CAPA-IVM compared to conventional IVF after a longer follow-up period. Does the development between the two groups have a clinically significant difference? Based on these questions, we decided to conduct an assessment of the physical, behavioural, mental, and motor development of children born from CAPA-IVM and conventional IVF up to 5 years after birth.

ELIGIBILITY:
Inclusion Criteria:

* All babies born following the In-vitro Maturation and In-vitro fertilization from our FM study (NCT03405701) participated in our previous follow-up study (NCT04296357)
* Parents agree to participate in the study.

Exclusion Criteria:

* Babies died under or at 60 months

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children participated in our previous follow-up study (NCT04296357)
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Normal ASQ-3 score rate. | Up to 5 years after birth
  A normal ASQ-3 score is the child's total score for each area above the cutoff. ASQ-3 (Ages and Stages Questionaires®) has 5 aspects: Communication, Gross motor, Fine motor, Problem solving, and Personal-Social Each aspect has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. ASQ-3 score = total area scores.
Normal SDQ score rate. | Up to 5 years after birth
  Normal SDQ score is defined as the total score of each area out of the abnormal range for each one.
  Abnormal range for each area is described as below:
  1. emotional symptoms: from 5 to 10
  2. conduct problems: from 4 to 10
  3. hyperactivity/inattention: from 7 to 10
  4. peer relationship problems: from 4 to 10
  5. prosocial behaviour: from 0 to 4
  6. The total difficulties score: from 17 to 40
Normal weight rate | Up to 5 years after birth
  Normal weight is a BMI greater than or equal to -2 standard deviations and less than or equal to 1 standard deviation of the WHO growth reference median.

SECONDARY OUTCOMES:
Thinness rate | Up to 5 years after birth
  Thinness is a BMI less than -2 standard deviations below the WHO growth reference median.
Overweight rate | Up to 5 years after birth
  Overweight is a BMI greater than 1 standard deviations above the WHO growth reference median.
Obesity rate | Up to 5 years after birth
  Obesity is a weight greater than 2 standard deviations above the WHO growth reference median.
Score of Communication (ASQ-3 questionnaire) | Up to 5 years after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Gross motor (ASQ-3 questionnaire) | Up to 5 years after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Fine motor (ASQ-3 questionnaire) | Up to 5 years after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Problem solving (ASQ-3 questionnaire) | Up to 5 years after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Personal-Social (ASQ-3 questionnaire) | Up to 5 years after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspect in each stage has an alternative threshold.
Score of Emotional symptoms (SDQ questionnaire) | Up to 5 years after birth
  5 questions, if the answer is Not True, score = 0, Somewhat True = 1 and Certianly True = 2.
  Normal SDQ score is defined as the total score of each area out of the abnormal range for each one.
  The abnormal range for Emotional symptoms is from 5 to 10.
Score of Conduct problems (SDQ questionnaire) | Up to 5 years after birth
  5 questions, if the answer is Not True, score = 0, Somewhat True = 1 and Certianly True = 2.
  This area has a question: "Generally well behaved, usually does what adults request." It needs to change the score to Not True, score = 2, Somewhat True = 1, and Certainly True = 0.
  Normal SDQ score is defined as the total score of each area out of the abnormal range for each one.
  Abnormal range for Conduct problems is from 4 to 10.
Score of hyperactivity/inattention (SDQ questionnaire) | Up to 5 years after birth
  5 questions, if the answer is Not True, score = 0, Somewhat True = 1 and Certianly True = 2.
  This area has two questions: "Thinks things out before acting" and "Good attention span, sees work through to the end." They need to change the score to Not True, score = 2, Somewhat True = 1, and Certainly True = 0.
  Normal SDQ score is defined as the total score of each area out of the abnormal range for each one.
  Abnormal range for hyperactivity/inattention is from 8 to 10.
Score of peer relationship problems (SDQ questionnaire) | Up to 5 years after birth
  5 questions, if the answer is Not True, score = 0, Somewhat True = 1 and Certianly True = 2.
  This area has two questions: "Has at least one good friend?" and "Generally liked by other children. "They need to change the scores to Not True, score = 2, Somewhat True, score = 1, and Certainly True, score = 0.
  Normal SDQ score is defined as the total score of each area out of the abnormal range for each one.
  Abnormal range for peer relationship problems is from 4 to 10.
Score of prosocial behavior (SDQ questionnaire) | Up to 5 years after birth
  5 questions, if the answer is Not True, score = 0, Somewhat True = 1 and Certianly True = 2.
  Normal SDQ score is defined as the total score of each area out of the abnormal range for each one.
  Abnormal range for prosocial behavior is from 0 to 6.
The total difficulties score. | Up to 5 years after birth
  The total difficulties score is generated by adding the score of emotional symptoms, conduct problems, hyperactivity/inattention and peer relationship problems together.
  The abnormal range for the total difficulties score is from 17 to 40.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No